CLINICAL TRIAL: NCT03922139
Title: OnabotulinumtoxinA (Botox) Effect on Pain and Return to Sport in Chronic Exertional Compartment Syndrome of the Anterior Leg: A Pilot Study
Brief Title: Botox for the Treatment of Chronic Exertional Compartment Syndrome
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: due to COVID-19
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1061; Ortho Rehab (Other: UW Madison); Protocol Version 6/15/2020 (Other: UW Madison); A536760 (Other: UW Madison); SMPH\PEDIATRICS\GPAM (Other: UW Madison)
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Results first posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Compartment Syndrome of Leg
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Botox (Experimental): Ultrasound guided 1 mg/1 mL injection.
  25 units of Botox will be injected 2 cm proximal and 2 cm distal to the midpoint of the tibialis anterior muscle.
  Interventions: Drug: OnabotulinumtoxinA Injection

INTERVENTIONS:
Drug: OnabotulinumtoxinA Injection — Ultrasound guided 1 mg/1 mL injection.
  25 units of Botox will be injected 2 cm proximal and 2 cm distal to the midpoint of the tibialis anterior muscle.
  Other Names: Botox

SUMMARY:
After diagnosis of Chronic Exertional Compartment Syndrome (CECS), the participants will be referred to both physical therapy and Botox injection. In physical therapy, the therapist will perform strength measurements of the lower leg (ankle plantarflexion and dorsiflexion) which will be repeated 2 months following the injection. An ultrasound-guided injection of 50 units of Botox will be administered into the tibialis anterior. 25 units will be injected into two different spots in the muscle one being more proximal and the other distal. This will be a one-time injection and will be observed as to how it effects participant symptoms over the next 6 months at either a clinic visit (at 2 months) or telephone call (at 4 and 6 months after injection) via the University of Wisconsin Running Index. Two months following the injection, the participant will undergo repeat measurements of strength using the Kiio Force Sensor.

Should potential participants of childbearing potential wish to enroll in the study, a urine pregnancy test will be performed prior to enrollment; participants will not be enrolled if test is positive.

DETAILED DESCRIPTION:
Chronic exertional compartment syndrome (CECS) is an overuse injury first described by Mavor in 1956 that typically affects young endurance athletes, classically distance runners. CECS occurs primarily in the lower leg, predominantly in the anterior compartment, although it has been reported elsewhere in the body.

The pathophysiology of CECS is not completely understood. Similar to acute compartment syndrome, it is thought to result from increased pressure within the restrictions of the fascial planes of a muscle compartment. Exercise increases blood flow to active muscles causing them to expand. If constricted by surrounding noncompliant fascia, such swelling increases pressure within the muscle compartment. Ultimately, pressure within the compartment reduces blood flow leading to muscle ischemia and pain when metabolic demands cannot be met. Several studies have demonstrated decreased blood flow and oxygenation in the legs of symptomatic patients with CECS.

Cessation of inciting activities resolves symptoms in most cases of CECS. Without this cessation, the prognosis for CECS is poor if treated non-operatively. Should symptoms continue, patients are referred for possible muscle compartment release, currently the most widely accepted treatment approach despite a significant number of treatment failures. To date, no alternative non-operative approach has successfully treated refractory symptoms.

Recently, it has been hypothesized that botulinum toxin could reduce intramuscular pressure in CECS . Isner-Horoboti et al, performed abobotulinum toxin A injections into the anterior and anterior/lateral compartments in 16 individuals with a mean follow up of 4.4 months (range 3-6 months). Fifteen (95%) patients were asymptomatic after intervention with fourteen (88%) exhibiting normalized post-exercise compartment pressures. Using manual muscle testing, they determined that 11 patients displayed decreased strength though did not produce noticeable subjective weakness. A later case report by Baria and Sellon presented the first long-term follow up (14 months) of a CECS case treated with botulinum toxin injections (Botox) in which the patient reported continued pain relief and had resumed her active lifestyle without adverse effects.

The proposed investigation will aim to build upon the results of existing studies. The novelty of this approach involves a differing dosage of the toxin (Botox) into a more targeted muscle group, specifically the tibialis anterior, while also utilizing a smaller dosage than in previous studies. Further, while previous studies have used manual muscle testing to test strength, many studies have found this method unreliable. As such, a Kiio force sensor will be used at multiple time points to determine weakness quantitatively. Lastly, the reliable and validated University of Wisconsin Running Index will be used to evaluate return to sport.

After diagnosis of CECS, the participants will be referred to both physical therapy and Botox injection. In physical therapy, the therapist will perform strength measurements of the lower leg (ankle plantarflexion and dorsiflexion) which will be repeated 2 months following the injection. An ultrasound-guided injection of 50 units of Botox into the tibialis anterior will be performed. 25 units will be injected into two different spots in the muscle, one being more proximal and the other distal. This will be a one-time injection that will be monitored to see how it effects participant symptoms over the next 6 months at either a clinic visit (at 2 months) or telephone call (at 4 and 6 months after injection) via the University of Wisconsin Running Index. Two months following the injection, the participant will undergo repeat measurements of strength using the Kiio Force Sensor.

Should potential participants be of childbearing potential wish to enroll in the study, a urine pregnancy test will be performed prior to enrollment; participants will not be enrolled if test is positive.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written informed consent
* Willing to comply with all study procedures and be available for the duration of the study including reliable use of telephone for communication
* Male or female, at least 18 years of age
* Documented diagnosis of CECS
* Females of childbearing potential must have a negative urine pregnancy test prior to enrollment and agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to enrollment and for the duration of study participation. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: Has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Be involved, either competitively or non-competitively, in an activity requiring significant running as determined by the PI

Exclusion Criteria:

* History of hypersensitivity or allergy to any of the study drugs or drugs of similar chemical classes
* Known neuromuscular disease
* Known pulmonary disease including but not limited to asthma, pneumonia, or upper respiratory tract infection
* Dysphagia
* Known cardiac disease including but not limited to congestive heart failure, arrhythmia, or history of myocardial infarction
* History of lower extremity fasciotomy
* Enrolled in another clinical trial or has used any investigational drugs, biologics, or devices within 30 days prior to enrollment
* Currently or have taken in the past medications that affect neuromuscular function: aminoglycosides, muscle relaxants, or other botulinum neurotoxin agents
* Women who are pregnant or breast-feeding
* Vulnerable populations
* Not suitable for study participation due to other reasons at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Suer, MD, Principal Investigator — UW Madison - SMPH, Department of Orthopedics and Rehabilitation
Locations (1):
- Pain Management Clinic, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the University of Wisconsin - Madison from October 2019 to February 2021.
Groups:
- Botox: Ultrasound guided 1 mg/1 mL injection.
  25 units of Botox will be injected 2 cm proximal and 2 cm distal to the midpoint of the tibialis anterior muscle.
  OnabotulinumtoxinA Injection: Ultrasound guided 1 mg/1 mL injection.
  25 units of Botox will be injected 2 cm proximal and 2 cm distal to the midpoint of the tibialis anterior muscle.
Period: Overall Study
Arm/Group | Botox
Started | 7
Completed 2 Month Surveys | 7
Completed 4 Month Surveys | 6
Completed 6 Month Surveys | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Botox
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Relief of Pain
Description: Percentage of Relief of Pain will be assessed at each time point (2,4,6 months) using Friedman's ANOVA.
Time Frame: Baseline, 2 months, 4 months and 6 months
Population: not all participants completed the assessment for all time points
Measure: Mean (Full Range); unit: percentage relief of pain
Arm/Group | Botox
Number analyzed (Participants) | 7
percentage relief of pain
  Baseline | 0 [0 to 0]
  2 months | 80.7 [0 to 100]
  4 months: number analyzed (Participants) | 5
  4 months | 100 [100 to 100]
  6 months: number analyzed (Participants) | 6
  6 months | 100 [100 to 100]

2. Primary Outcome: Number of Participants With Lower Extremity Weakness
Description: A primary safety endpoint is the incidence of lower extremity weakness
Time Frame: up to 6 months
Population: one participant dropped from the study
Measure: Count of Participants; unit: Participants
Arm/Group | Botox
Number analyzed (Participants) | 6
Participants | 0

3. Primary Outcome: Incidence of Adverse Events
Description: A primary safety endpoint is the incidence of adverse events, such as bruising, bleeding, pain, redness, or swelling where the injection was given.
Time Frame: up to 6 months
Measure: Number; unit: number of adverse events
Arm/Group | Botox
Number analyzed (Participants) | 7
number of adverse events | 0

4. Secondary Outcome: Change in Ankle Dorisflexsion Strength Using Kiio Force Sensor
Description: A Kiio Force Sensor will be used to measure the change in ankle strength. Change in strength outcomes at baseline and 2 months will be assessed using Wilcoxon signed rank tests or, if necessary, linear mixed effects models for repeated measures, to account for intra-subject correlation (left and right legs).
Time Frame: baseline and month 2
Population: one participant did not return for 2 month measures
Measure: Mean (Full Range); unit: degrees
Arm/Group | Botox
Number analyzed (Participants) | 7
degrees
  baseline left ankle | 24.6 [22.8 to 27.1]
  baseline right ankle | 24.6 [22.9 to 26.9]
  2 months left ankle: number analyzed (Participants) | 6
  2 months left ankle | 25.2 [23.5 to 27.3]
  2 months right ankle: number analyzed (Participants) | 6
  2 months right ankle | 25.0 [23.4 to 27.1]

5. Secondary Outcome: Change in Ankle Plantarflexion Strength Using Kiio Force Sensor
Description: as for outcome 4
Time Frame: baseline and month 2
Population: one participant did not return for 2 month measures
Measure: Mean (Full Range); unit: degrees
Arm/Group | Botox
Number analyzed (Participants) | 7
degrees
  baseline left ankle | 172.5 [158.1 to 190.1]
  baseline right ankle | 173.8 [158.4 to 192.0]
  2 months left ankle: number analyzed (Participants) | 6
  2 months left ankle | 176.5 [162.1 to 191.8]
  2 months right ankle: number analyzed (Participants) | 6
  2 months right ankle | 177.0 [162.4 to 192.6]

6. Secondary Outcome: Change in Ankle Inversion Strength Using Kiio Force Sensor
Description: as for outcome 4
Time Frame: baseline and month 2
Population: one participant did not return for 2 month measures
Measure: Mean (Full Range); unit: degrees
Arm/Group | Botox
Number analyzed (Participants) | 7
degrees
  Baseline left ankle | 22.4 [20.8 to 25.0]
  baseline right ankle | 22.6 [21.0 to 24.9]
  2 months left ankle: number analyzed (Participants) | 6
  2 months left ankle | 22.9 [21.8 to 25.2]
  2 months right ankle: number analyzed (Participants) | 6
  2 months right ankle | 23.1 [21.9 to 25.0]

7. Secondary Outcome: Change in Ankle Eversion Strength Using Kiio Force Sensor
Description: as for outcome 4
Time Frame: baseline and month 2
Population: one participant did not return for 2 month measures
Measure: Mean (Full Range); unit: degrees
Arm/Group | Botox
Number analyzed (Participants) | 7
degrees
  baseline left ankle | 22.8 [20.9 to 25.2]
  baseline right ankle | 22.7 [20.9 to 25.3]
  2 months left ankle: number analyzed (Participants) | 6
  2 months left ankle | 23.3 [21.0 to 25.4]
  2 months right ankle: number analyzed (Participants) | 6
  2 months right ankle | 23.3 [21.2 to 25.5]

8. Secondary Outcome: Change in Ability to Perform Activities of Daily Living
Description: A question on the UWRI asks the participant to indicate how their running injury impacts their ability to perform daily activities: No Impact, Slightly Impact, Moderately Impact, Significantly Impact, Unable to Perform.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: One participant did not answer the 4 month survey
Measure: Count of Participants; unit: Participants
Arm/Group | Botox
Number analyzed (Participants) | 7
Participants
  baseline: No Impact | 2
  baseline: Slightly Impact | 0
  baseline: Moderately Impact | 2
  baseline: Significantly Impact | 3
  baseline: Unable to Perform | 0
  2 months: No Impact | 4
  2 months: Slightly Impact | 3
  2 months: Moderately Impact | 0
  2 months: Significantly Impact | 0
  2 months: Unable to Perform | 0
  4 months: number analyzed (Participants) | 6
  4 months: No Impact | 6
  4 months: Slightly Impact | 0
  4 months: Moderately Impact | 0
  4 months: Significantly Impact | 0
  4 months: Unable to Perform | 0
  6 months: No Impact | 7
  6 months: Slightly Impact | 0
  6 months: Moderately Impact | 0
  6 months: Significantly Impact | 0
  6 months: Unable to Perform | 0

9. Secondary Outcome: Participant Frustration With Injury
Description: A question on the UWRI asks the participant to indicate how frustrated they are by their running injury: Not frustrated, Mildly frustrated, Moderately frustrated, Significantly frustrated, or Extremely frustrated.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: one participant did not answer 4 month survey
Measure: Count of Participants; unit: Participants
Arm/Group | Botox
Number analyzed (Participants) | 7
Participants
  baseline: Not Frustrated | 0
  baseline: Mildly Frustrated | 1
  baseline: Moderately Frustrated | 1
  baseline: Significantly Frustrated | 1
  baseline: Extremely Frustrated | 4
  2 months: Not Frustrated | 5
  2 months: Mildly Frustrated | 2
  2 months: Moderately Frustrated | 0
  2 months: Significantly Frustrated | 0
  2 months: Extremely Frustrated | 0
  4 months: number analyzed (Participants) | 6
  4 months: Not Frustrated | 5
  4 months: Mildly Frustrated | 1
  4 months: Moderately Frustrated | 0
  4 months: Significantly Frustrated | 0
  4 months: Extremely Frustrated | 0
  6 months: Not Frustrated | 7
  6 months: Mildly Frustrated | 0
  6 months: Moderately Frustrated | 0
  6 months: Significantly Frustrated | 0
  6 months: Extremely Frustrated | 0

10. Secondary Outcome: Participant Perception of Recovery From Injury
Description: A question on the UWRI asks the participant to indicate how much recovery have they made from their running injury: Complete Recovery, Significant Recovery, Moderate Recovery, Minimal Recovery, No Recovery.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: One participant did not answer the 4 month survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Botox
Number analyzed (Participants) | 7
Participants
  baseline: Complete Recovery | 0
  baseline: Significant Recovery | 0
  baseline: Moderate Recovery | 1
  baseline: Minimal Recovery | 1
  baseline: No Recovery | 5
  2 months: Complete Recovery | 3
  2 months: Significant Recovery | 4
  2 months: Moderate Recovery | 0
  2 months: Minimal Recovery | 0
  2 months: No Recovery | 0
  4 months: number analyzed (Participants) | 6
  4 months: Complete Recovery | 5
  4 months: Significant Recovery | 1
  4 months: Moderate Recovery | 0
  4 months: Minimal Recovery | 0
  4 months: No Recovery | 0
  6 months: Complete Recovery | 7
  6 months: Significant Recovery | 0
  6 months: Moderate Recovery | 0
  6 months: Minimal Recovery | 0
  6 months: No Recovery | 0

11. Secondary Outcome: Pain in the 24 Hours Following Running
Description: A question on the UWRI asks the participant to indicate how much pain they experience during the 24 hours following a run: No pain, Minimal pain, Moderate pain, Significant pain, Unable to Run.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: One participant did not complete the 4 month survey
Measure: Count of Participants; unit: Participants
Arm/Group | Botox
Number analyzed (Participants) | 7
Participants
  baseline: No Pain | 2
  baseline: Minimal Pain | 3
  baseline: Moderate Pain | 1
  baseline: Significant Pain | 0
  baseline: Unable to Run | 1
  2 months: No Pain | 7
  2 months: Minimal Pain | 0
  2 months: Moderate Pain | 0
  2 months: Significant Pain | 0
  2 months: Unable to Run | 0
  4 months: number analyzed (Participants) | 6
  4 months: No Pain | 6
  4 months: Minimal Pain | 0
  4 months: Moderate Pain | 0
  4 months: Significant Pain | 0
  4 months: Unable to Run | 0
  6 months: No Pain | 7
  6 months: Minimal Pain | 0
  6 months: Moderate Pain | 0
  6 months: Significant Pain | 0
  6 months: Unable to Run | 0

12. Secondary Outcome: Change in Running Duration: Weekly
Description: A question on the UWRI asks the participant to indicate if their weekly mileage or weekly running time changed as a result of their injury: Same or greater than before injury, Minimally reduced, Moderately reduced, Significantly reduced, Unable to Run.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: One participant did not complete the 4 month survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Botox
Number analyzed (Participants) | 7
Participants
  baseline: Same or greater than before injury | 0
  baseline: Minimally reduced | 0
  baseline: Moderately reduced | 2
  baseline: Significantly reduced | 3
  baseline: Unable to Run | 2
  2 months: Same or greater than before injury | 6
  2 months: Minimally reduced | 1
  2 months: Moderately reduced | 0
  2 months: Significantly reduced | 0
  2 months: Unable to Run | 0
  4 months: number analyzed (Participants) | 6
  4 months: Same or greater than before injury | 6
  4 months: Minimally reduced | 0
  4 months: Moderately reduced | 0
  4 months: Significantly reduced | 0
  4 months: Unable to Run | 0
  6 months: Same or greater than before injury | 7
  6 months: Minimally reduced | 0
  6 months: Moderately reduced | 0
  6 months: Significantly reduced | 0
  6 months: Unable to Run | 0

13. Secondary Outcome: Change in Running Duration: Longest Run
Description: A question on the UWRI asks the participant to indicate if the distance of their longest weekly run has changed as a result of their injury: Same or longer than before my injury, Minimally reduced, Moderately reduced, Significantly reduced, Unable to Run.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: One participant did not complete the 4 month survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Botox
Number analyzed (Participants) | 7
Participants
  baseline: Same or longer than before my injury | 1
  baseline: Minimally reduced | 0
  baseline: Moderately reduced | 2
  baseline: Significantly reduced | 4
  baseline: Unable to Run | 0
  2 months: Same or longer than before my injury | 6
  2 months: Minimally reduced | 1
  2 months: Moderately reduced | 0
  2 months: Significantly reduced | 0
  2 months: Unable to Run | 0
  4 months: number analyzed (Participants) | 6
  4 months: Same or longer than before my injury | 6
  4 months: Minimally reduced | 0
  4 months: Moderately reduced | 0
  4 months: Significantly reduced | 0
  4 months: Unable to Run | 0
  6 months: Same or longer than before my injury | 7
  6 months: Minimally reduced | 0
  6 months: Moderately reduced | 0
  6 months: Significantly reduced | 0
  6 months: Unable to Run | 0

14. Secondary Outcome: Change in Running Speed
Description: A question on the UWRI asks the participant to indicate if the distance of the longest weekly run has changed as a result of their injury: Same or faster than before my injury, Minimally reduced, Moderately reduced, Significantly reduced, Unable to Run.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: One participant did not complete the 4 month survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Botox
Number analyzed (Participants) | 7
Participants
  baseline: Same or faster than before my injury | 0
  baseline: Minimally reduced | 2
  baseline: Moderately reduced | 1
  baseline: Significantly reduced | 2
  baseline: Unable to Run | 2
  2 months: Same or faster than before my injury | 7
  2 months: Minimally reduced | 0
  2 months: Moderately reduced | 0
  2 months: Significantly reduced | 0
  2 months: Unable to Run | 0
  4 months: number analyzed (Participants) | 6
  4 months: Same or faster than before my injury | 6
  4 months: Minimally reduced | 0
  4 months: Moderately reduced | 0
  4 months: Significantly reduced | 0
  4 months: Unable to Run | 0
  6 months: Same or faster than before my injury | 7
  6 months: Minimally reduced | 0
  6 months: Moderately reduced | 0
  6 months: Significantly reduced | 0
  6 months: Unable to Run | 0

15. Secondary Outcome: Participant Confidence in Increasing the Duration and Intensity of Running
Description: A question on the UWRI asks the participant to indicate how their injury affects their confidence to increase the duration or intensity of their running: Confident to increase my running, If I increase I might be fine, Neutral, If I increase I might get worse, I cannot increase my running.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: One participant did not complete the 4 month survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Botox
Number analyzed (Participants) | 7
Participants
  baseline: Confident to increase my running | 1
  baseline: If I increase I might be fine | 0
  baseline: Neutral | 0
  baseline: If I increase I might get worse | 3
  baseline: I cannot increase my running | 3
  2 months: Confident to increase my running | 5
  2 months: If I increase I might be fine | 1
  2 months: Neutral | 1
  2 months: If I increase I might get worse | 0
  2 months: I cannot increase my running | 0
  4 months: number analyzed (Participants) | 6
  4 months: Confident to increase my running | 6
  4 months: If I increase I might be fine | 0
  4 months: Neutral | 0
  4 months: If I increase I might get worse | 0
  4 months: I cannot increase my running | 0
  6 months: Confident to increase my running | 7
  6 months: If I increase I might be fine | 0
  6 months: Neutral | 0
  6 months: If I increase I might get worse | 0
  6 months: I cannot increase my running | 0

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | Botox
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT03922139/Prot_SAP_000.pdf